CLINICAL TRIAL: NCT02487511
Title: Comparison of the Eradication Rate Between 1- and 2-Week PPI Containing Therapies for Helicobacter Pylori Eradication
Brief Title: Eradication Rate Between 1- and 2-Week Helicobacter Pylori Eradication Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St.Paul's Hospital, Korea (Other)
Responsible Party: Principal Investigator, JUNG HWAN OH, Associate Professor, St.Paul's Hospital, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HPTX Duration
Record Dates: First submitted 2015-06-25; First posted 2015-07-01 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: H.Pylori Gastrointestinal Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 14 days (Active Comparator): 14 days treatment regimen
  Interventions: Other: Duration of HP therapy
- 7 days (No Intervention): 7 days treatment regimen

INTERVENTIONS:
Other: Duration of HP therapy — the comparison of HP eradication rate between 7 days and 14 days
  Arms: 14 days

SUMMARY:
It is recommended as the first line treatment regimen to eradicate Helicobacter pylori (HP), 7 or 14 days treatment of proton pump inhibitor (PPI) based triple therapy consisting of one PPI and two antibiotics, clarithromycin and amoxicillin. In the case of treatment failure, 7 or 14 days of quadruple therapy (PPI＋metronidazole＋tetracycline＋bismuth) is recommended.

This study aims to investigate which duration would be better for eradication of HP. The study design is a randomized controlled trial. The patients were randomly assigned to 7 days or 14 days treatment groups. Primary endpoint was the eradication rate of PPI based triple therapy. Secondary endpoints were to compare the rate of drug compliance and side effects in both groups.

DETAILED DESCRIPTION:
The recommended duration of triple therapy is typically 10 to 14 days in the United States and 7 days in Europe. In Korea, it is recommended as the first line treatment regimen, 7 or 14 days treatment of proton pump inhibitor (PPI) based triple therapy consisting of one PPI and two antibiotics, clarithromycin and amoxicillin. In case for treatment failure which is often related to Helicobacter pylori (HP) resistance to clarithromycin or metronidazole, bismuth-based quadruple therapy is commonly used as second-line therapy, however, the eradication rates was widely ranged according to the treatment duration.

The objective of the study is to investigate whether treatment duration would affect the eradication rate of HP as a PPI based triple therapy (1st line therapy) and a bismuth-based quadruple therapy (2nd line therapy).

ELIGIBILITY:
Inclusion Criteria:

* Peptic ulcer including ulcer scar
* Early gastric cancer
* Gastric mucosa-associated lymphoid tissue lymphoma

Exclusion Criteria:

* operation history
* liver cirrhosis
* chronic kidney disease
* pregnancy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
the comparison with 7days and 14days eradication rate of PPI based therapy | 12 months after randomization

SECONDARY OUTCOMES:
the rate of side effects related to helicobacter eradication regimen | 12 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: JUNG HWAN Oh, MD, PhD, Principal Investigator — the Catholic Univerisity of Korea
Locations (1):
- The Catholic University of Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim TH, Park JM, Cheung DY, Oh JH. Comparison of 7- and 14-Day Eradication Therapy for Helicobacter pylori with First- and Second-Line Regimen: Randomized Clinical Trial. J Korean Med Sci. 2020 Feb 10;35(5):e33. doi: 10.3346/jkms.2020.35.e33. PMID 32030921